CLINICAL TRIAL: NCT03675581
Title: A Phase I Trial to Investigate the Effect of Nintedanib on the Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Female Patients With Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Brief Title: A Study to Test Whether Nintedanib Influences the Components of Birth-control Pills in Women With Systemic Sclerosis Associated Interstitial Lung Disease (SSc-ILD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0340; 2018-001177-24 (EudraCT Number)
Record Dates: First submitted 2018-09-17; First posted 2018-09-18 (Actual); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Scleroderma, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — ethinyl estradiol, levonorgestrel drug combination; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental)
  Interventions: Drug: Microgynon; Drug: Nintedanib

INTERVENTIONS:
Drug: Microgynon — fixed sequence trial
Drug: Nintedanib — fixed sequence trial

SUMMARY:
The main objective is to assess the potential influence of continuous intake of nintedanib on the systemic exposure of ethinylestradiol and levonorgestrel when administered in combination.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* A woman of non-child bearing potential, i.e. being postmenopausal1 or permanently sterilised (e.g. hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or a woman of childbearing potential correctly and consistently using a highly effective method of non-hormonal birth control (i.e. IUD or bilateral tubal ligation) together with barrier methods at least 30 days prior to first administration of Microgynon® (Visit 2), during the trial and for 3 months after last intake of nintedanib.
* 2013 American College of Rheumatology (ACR) / European League against Rheumatism (EULAR) classification criteria for Systemic Sclerosis associated Interstitial Lung Disease (SSc) fulfilled
* SSc related Interstitial Lung Disease confirmed by High Resolution Computer Tomography (HRCT); Extent of fibrotic disease in the lung >= 10%
* Forced Vital Capacity (FVC) >= 40% of predicted normal
* Carbon Monoxide Diffusion Capacity (DLCO) 30% to 89% of predicted normal
* Further inclusion criteria apply

Exclusion criteria:

* Aspartate Transaminase (AST), Alanine Transaminase (ALT) >1.5 x Upper Level of Normal (ULN).
* Bilirubin >1.5 x ULN
* Creatinine clearance <30 mL/min
* Clinically relevant anaemia at investigators discretion
* Airway obstruction (pre-bronchodilator Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) <0.7)
* Other clinically significant pulmonary abnormalities
* Significant Pulmonary Hypertension (PH)
* Cardiovascular diseases
* More than 3 digital fingertip ulcers or a history of severe digital necrosis requiring hospitalization or severe other ulcers
* Bleeding risk (such as predisposition to bleeding, fibrinolysis, full-dose anticoagulation, high dose antiplatelet therapy, history of hemorrhagic central nervous system (CNS) event within last year
* International normalised ratio (INR) >2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by >1.5 x ULN)
* History of thrombo-embolic event within last year
* Previous or planned hematopoietic stem cell transplantation
* Clinical signs of malabsorption or needing parenteral nutrition
* Patients with underlying chronic liver disease (Child Pugh A, B, C hepatic impairment)
* Previous treatment with nintedanib or pirfenidone
* Further exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- UNIV UZ Gent, Ghent, Belgium
- France (2):
  - HOP Avicenne, Bobigny
  - HOP Bichat, Paris
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Portugal (2):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Fernando Fonseca, EPE, Amadora
- Spain (2):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.

REFERENCES:
- [Derived] Vonk MC, Guillen-Del-Castillo A, Kreuter M, Avis M, Marzin K, Mack SR, Wind S, Gahlemann M. A Drug-Drug Interaction Study to Investigate the Effect of Nintedanib on the Pharmacokinetics of Microgynon (Ethinylestradiol and Levonorgestrel) in Female Patients with Systemic Sclerosis-Associated Interstitial Lung Disease. Eur J Drug Metab Pharmacokinet. 2022 Jan;47(1):81-89. doi: 10.1007/s13318-021-00728-7. Epub 2021 Oct 18. PMID 34664183
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an open-label, 2-period, fixed-sequence, Phase I trial in order to investigate the effect of nintedanib on the pharmacokinetics of a combination of ethinylestradiol and levonorgestrel in female patients with Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD).
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. Patients attended a specialist site which ensured that they (the patients) strictly met all inclusion and none of the exclusion criteria. Patients were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Microgynon / Microgynon + Nintedanib: Period 1 consisted of a Microgynon alone treatment. All patients received a single dose of Microgynon: 1 tablet of 30 μg ethinylestradiol and 150 μg levonorgestrel at trial Day -3 (Reference treatment, R).
  Period 2 consisted of a Microgynon + nintedanib combination treatment. All patients received a continuous stable dose of nintedanib, soft gelatine capsule of 150 milligrams (mg) twice daily (bid) (300 mg total per day), starting from trial Day 1 over a period of at least 14 days to approximately 28 days. After at least 10 days of nintedanib treatment, all patients received a second single dose of Microgynon: 1 tablet of 30 μg ethinylestradiol and 150 μg levonorgestrel on trial Day 11 (Test treatment, T).
  All treatments were to be taken with food, swallowed whole with approximately 250 milliliters (mL) of water and was not to be chewed or crushed.
Period: Period 1: Microgynon Alone
Arm/Group | Microgynon / Microgynon + Nintedanib
Started | 17
Completed | 17
Not Completed | 0
Period: Period 2: Microgynon + Nintedanib
Arm/Group | Microgynon / Microgynon + Nintedanib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Arm/Group | Microgynon / Microgynon + Nintedanib
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of Ethinylestradiol in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of ethinylestradiol in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of ethinylestradiol were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after microgynon administration alone or in combination with nintedanib.
Population: Pharmacokinetic parameter analysis set (PKS): The PKS included all subjects in the treated set (TS) who provided at least 1 pharmacokinetic (PK) endpoint that had been defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Standard Error); unit: picograms * hours per milliliters
Groups:
- Microgynon Alone (Reference Treatment, R): Period 1 consisted of a Microgynon alone treatment. All patients received a single dose of Microgynon: 1 tablet of 30 μg ethinylestradiol and 150 μg levonorgestrel at trial Day -3 (Reference treatment, R).
  The treatment was to be taken with food, swallowed whole with approximately 250 milliliters (mL) of water and was not to be chewed or crushed.
- Microgynon + Nintedanib (Test Treatment, T): Period 2 consisted of a Microgynon + nintedanib combination treatment. All patients received a continuous stable dose of nintedanib, soft gelatine capsule of 150 milligrams (mg) twice daily (bid) (300 mg total per day), starting from trial Day 1 over a period of at least 14 days to approximately 28 days. After at least 10 days of nintedanib treatment, all patients received a second single dose of Microgynon: 1 tablet of 30 μg ethinylestradiol and 150 μg levonorgestrel on trial Day 11 (Test treatment, T).
  The treatment was to be taken with food, swallowed whole with approximately 250 milliliters (mL) of water and was not to be chewed or crushed.
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms * hours per milliliters | 610.00 (1.16) | 618.28 (1.16)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; The statistical model was analysis of variance (ANOVA) on the logarithmic scale considering the effects "subjects" as random and "treatment" as fixed; Ratio of the geometric means (T/R) % = 101.36, 90% CI 2-sided [92.83 to 110.67], Standard Deviation 13.7 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

2. Primary Outcome: Area Under the Concentration-time Curve of Levonorgestrel in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of levonorgestrel in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
  For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of levonorgestrel were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms * hours per milliliters
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms * hours per milliliters | 33062.73 (1.20) | 31872.47 (1.20)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 96.40, 90% CI 2-sided [91.48 to 101.58], Standard Deviation 8.2 — The standard deviation is actually the geometric coefficient of variation (gCV) T = Test, R = Reference

3. Primary Outcome: Maximum Measured Concentration of Ethinylestradiol in Plasma (Cmax)
Description: Maximum measured concentration of ethinylestradiol in plasma (Cmax). For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of ethinylestradiol were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms per milliliters
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms per milliliters | 54.75 (1.11) | 63.89 (1.11)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 116.69, 90% CI 2-sided [107.63 to 126.51], Standard Deviation 12.6 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

4. Primary Outcome: Maximum Measured Concentration of Levonorgestrel in Plasma (Cmax)
Description: Maximum measured concentration of levonorgestrel in plasma (Cmax). For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of levonorgestrel were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms per milliliters
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms per milliliters | 3124.48 (1.14) | 3152.35 (1.14)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 100.89, 90% CI 2-sided [89.90 to 113.23], Standard Deviation 18.1 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

5. Secondary Outcome: Area Under the Concentration-time Curve of Ethinylestradiol in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of ethinylestradiol in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of ethinylestradiol were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms * hours per milliliters
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms * hours per milliliters | 749.65 (1.14) | 758.95 (1.14)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 101.24, 90% CI 2-sided [93.95 to 109.10], Standard Deviation 11.7 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

6. Secondary Outcome: Area Under the Concentration-time Curve of Levonorgestrel in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of levonorgestrel in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  For Microgynon (ethinylestradiol + levonorgestrel) alone (Reference treatment, R) and Microgynon (ethinylestradiol + levonorgestrel) + nintedanib (Test treatment, T) plasma concentrations of levonorgestrel were measured 35 minutes (min) before and at 30 min, 1 hour (h), 1h 30 min, 2h, 3h, 4h, 6h, 8h, 11h 55 min, 23h 55 min, 47h 55 min after Microgynon administration alone or in combination with nintedanib.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms * hours per milliliters
Arm/Group | Microgynon Alone (Reference Treatment, R) | Microgynon + Nintedanib (Test Treatment, T)
Number analyzed (Participants) | 15 | 15
picograms * hours per milliliters | 56311.68 (1.24) | 49605.41 (1.24)
Statistical Analysis 1: Comparison: Microgynon Alone (Reference Treatment, R) vs Microgynon + Nintedanib (Test Treatment, T); Test type: Other — Relative systemic exposure; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of the geometric means (T/R) % = 88.09, 90% CI 2-sided [80.03 to 96.96], Standard Deviation 15.0 — The standard deviation is actually the geometric coefficient of variation (gCV) T=Test, R=Reference

ADVERSE EVENTS:
Time Frame: The adverse events collection time frame started at the day of first administration of the treatment till 2 days after for Microgynon alone, till 10 days after for nintedanib (before combination treatment), till 2 days after for Microgynon + nintedanib and as from 3 days after the combination treatment for nintedanib alone.
Description: Treated set (TS): The TS included all subjects who had been enrolled and treated with at least 1 dose of study drug. The treated set was used for safety analyses.
Groups:
- Nintedanib Alone (Before Combination Treatment): All patients received a continuous stable dose of nintedanib, 150 mg twice daily (bid) (300 mg total per day), soft gelatine capsule from trial Day 1 for at least 10 consecutive days.
  The treatment was to be taken with food, swallowed whole with approximately 250 mL of water and was not to be chewed or crushed.
- Microgynon + Nintedanib (Test Treatment, T): Period 2 consisted of a Microgynon + nintedanib combination treatment. All patients received a continuous stable dose of nintedanib, soft gelatine capsule of 150 milligrams (mg) twice daily (bid) (300 mg total per day), starting from trial Day 1 over a period of at least 14 days to approximately 28 days. After at least 10 days of nintedanib treatment, all patients received a second single dose of Microgynon: 1 tablet of 30 μg ethinylestradiol and 150 μg levonorgestrel on trial Day 11 (Test treatment, T).
  The treatment was to be taken with food, swallowed whole with approximately 250 mL of water and was not to be chewed or crushed.
- Nintedanib Alone (After Combination Treatment): All patients continued to receive a stable dose of nintedanib, 150 mg bid (300 mg total per day), soft gelatine capsule after the combination treatment on trial Days 12 and 13. The treatment was to be taken with food, swallowed whole with approximately 250 mL of water and was not to be chewed or crushed. AE's are considered to have occurred on nintedanib alone (after combination treatment) if occurring on Day 14 or later, i.e. at least 3 days after combination treatment.
Arm/Group | Microgynon Alone (Reference Treatment, R) | Nintedanib Alone (Before Combination Treatment) | Microgynon + Nintedanib (Test Treatment, T) | Nintedanib Alone (After Combination Treatment)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 1/17 | 0/17
Other Adverse Events (participants affected / at risk) | 3/17 | 11/17 | 3/17 | 2/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon Alone (Reference Treatment, R) (N=17) | Nintedanib Alone (Before Combination Treatment) (N=17) | Microgynon + Nintedanib (Test Treatment, T) (N=17) | Nintedanib Alone (After Combination Treatment) (N=17)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Microgynon Alone (Reference Treatment, R) (N=17) | Nintedanib Alone (Before Combination Treatment) (N=17) | Microgynon + Nintedanib (Test Treatment, T) (N=17) | Nintedanib Alone (After Combination Treatment) (N=17)
Nausea (Gastrointestinal disorders) | 0 | 6 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03675581/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03675581/SAP_001.pdf